CLINICAL TRIAL: NCT06599203
Title: Prognostic Factors in Children with Diabetic Ketoacidosis
Brief Title: Children with Diabetic Ketoacidosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Diaa Eldin Mahmoud sayed, 71515,Assiut, Assiut University
Other Study IDs: diabetic ketoacidosis
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the present work we aim to

1. Response to therapy, During the management of DKA, acid base status, glycemia, and serum electrolytes are measured frequently to monitor the efficacy of treatment, detect complications of DKA and its treatment, and to determine resolution of DKA.
2. Clinical complication like cerebral injury / cerebral edema , cognitive impairment , acute kidney injury , hypokalemia.
3. Severity of DKA

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is a life-threatening condition, especially in individuals with Type 1 diabetes. It arises from a severe insulin deficiency, resulting in elevated blood glucose levels . In reaction, the body begins metabolizing fat for energy

, which causes the production of ketones. Ketone buildup in the blood results in metabolic acidosis, which produces symptoms including extreme thirst, frequent urination, stomach discomfort, nausea, vomiting, disorientation, and breath that smells like fruit .A chronic autoimmune disease known as Type 1 Diabetes Mellitus (T1DM) is characterized by the eradication of insulin-producing beta cells in the pancreas. Although it may happen at any age, it often starts to manifest in childhood or adolescent . In T1DM, the immune system incorrectly targets and kills the beta cells, leading to little or nonexistent insulin production . The hormone insulin is essential for controlling blood glucose levels . Because of this, T1DM patients need lifelong insulin medication in order to survive. Excessive thirst, frequent urination, exhaustion, and an increased susceptibility to infections are all typical signs of T1DM . The treatment of T1DM entails routine blood glucose monitoring, the use of insulin pumps or injections, a balanced diet, routine physical exercise, and the management of additional risk factors for complications .DKA is diagnosed based on clinical presentation and biochemical abnormalities, including hyperglycemia (blood glucose >200 mg/dL), venous pH of <7.3 or serum bicarbonate less than 15, and the presence of ketones in the blood or urine. Ill patients with Type-1 DM should be evaluated for DKA, which can coexist with or be triggered by other acute illnesses (infection, trauma, etc.). There may be a history of polydipsia, polyuria, polyphagia (early), anorexia (late), weight loss, fatigue, or recurrent infection. Patients and parents may also report poor school performance, lack of concentration, altered mental status, and confusion as well.Patients with metabolic acidosis classically display rapid, deep breathing (Kussmaul respirations). The breath may have a fruity odor due to respiratory aceton elimination. Neurologic findings range from alert, to lethargic and drowsy, to comatose correlated with the extent of acidosis. In order to treat DKA and prevent life-threatening consequences, immediate medical intervention essential. DKA calls for intravenous fluids, insulin therapy, and correction of electrolyte imbalances. It is indeed crucial to study Diabetic Ketoacidosis (DKA), its incidence, and the features of hospital admissions in order to understand and improve the management of this condition . Delayed treatment altered sensorium , lower bicarbonate , lower pH , elevated urea , elevated creatinine , higher sodium levels at admission are significant risk factors for mortality among children with diabetic keto acidosis at initial presentation .Majority of these factors signify severe disease , and this could be aggravated by delay in recognition and treatment. Overall mortality among children presenting with DKA as the initial presentation in type 1 Diabetes mellitus is 12.8% . (14)

ELIGIBILITY:
Inclusion Criteria:

Hospitalized diabetic patients aged from 1 year to 16 years with diabetic ketoacidosis

Exclusion Criteria:

1. Other endocrine diseases as thyroid disease or pituitary disease
2. Severe Hepatic Dysfunction or Chronic Kidney Dysfunction: Patients with significant liver or kidney impairment were excluded from the study.
3. History of Malignant Tumor: The study did not include individuals with a previous history of any malignant tumor

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with type 1 DM with clinical presentation and biochemical abnormalities, including hyperglycemia (blood glucose200 mg/dL), venous pH less than7.3 or serum bicarbonate less than 15, and the presence of ketones in the blood or urine (12). Ill patients with Type-1 DM should be evaluated for DKA, which can coexist with or be triggered by other acute illnesses (infection, trauma, etc.). There may be a history of polydipsia, polyuria, polyphagia (early), anorexia (late), weight loss, fatigue, or recurrent infection.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Method | Baseline
  Full history taking in the form of personal history age ,sex ,demographics including residence and socioeconomic status , feeding history ,family history .
  complete physical examination including body temperature , respiratory rate heart rate , weight , skin color .
  laboratory investigations including random blood glucose , ketones in urine , arterial blood gases ,complete blood count , electrolytes , kidney function test , liver function test.
  They will be managed with standard care that include insulin, intravenous fluids, and appropriate supportive care. Serial assays of serum electrolytes, glucose, and blood pH were analyzed and correlated with clinical outcomes of either discharge to home or death.
Sample size | Baseline
  Based on determining the primary outcome variable, the estimated minimum required sample size is 130 patients. The sample size shall be calculated using Epi-info version 7 software based on the following hypothesis:
  The primary outcome variable correlates the final outcome in diabetic ketoacidosis with different confounding covariates such as demographic characteristics, clinical characteristics, and biochemical parameters at presentation.
  Based on previous studies (H Zayed 2016 ), the prevalence of DKA in Egypt was 17 % and based on the percentage confidence limits of 5% and a confidence level = 90%.
Determination of response to therapy and clinical complication of DKA | Baseline
  Response to therapy during the management of DKA is determined by measuring acid base status, glycemia, and serum electrolytes, venous PH, serum bicarbonate concentration HCO3(mmol/ml), anion gap AG and urine ketones frequently to monitor the efficacy of treatment, detect complications of DKA and its treatment, and to determine resolution of DKA.